CLINICAL TRIAL: NCT01148472
Title: A Double-blind, Randomised, Multicenter, Comparative Study of Escitalopram and Duloxetine in Outpatients With Major Depressive Disorder
Brief Title: Efficacy and Tolerability of Escitalopram and Duloxetine in Outpatients With Major Depressive Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: H. Lundbeck A/S, H. Lundbeck A/S
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10990; 2004-005069-39 (EudraCT Number)
Record Dates: First submitted 2010-06-17; First posted 2010-06-22 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Major Depressive Disorder
Keywords: Depressive disorder, major; Randomized controlled trials; Antidepressive agents
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Escitalopram; Dexetimide; Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Escitalopram (Experimental)
  Interventions: Drug: Escitalopram
- Duloxetine (Active Comparator)
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Escitalopram — 20mg once daily; orally
  Other Names: Cipralex, Lexapro
  Arms: Escitalopram
Drug: Duloxetine — 60mg once daily; orally
  Other Names: Cymbalta
  Arms: Duloxetine

SUMMARY:
The primary objective of this study was to compare the efficacy of escitalopram with that of duloxetine in outpatients with Major Depressive Disorder (MDD) after 24 weeks of treatment. The study hypothesis was that there were clinically important differences between the two drugs in terms of efficacy and adverse event profiles.

DETAILED DESCRIPTION:
Depression is a common mental disorder that presents with depressed mood, loss of interest or pleasure, disturbed sleep or appetite, low energy, feelings of guilt or low self-worth, and poor concentration. The lifetime prevalence of Major Depressive Disorder (MDD) in community samples is 10-25% for women and 5-12% for men. Depression may become chronic or recurrent and lead to substantial impairments in an individual's ability to take care of his or her everyday responsibilities. At its worst, depression may lead to suicide. Depression is recurrent in 75-80% of patients and becomes chronic in 15-20% of depressed patients.

The selective serotonin reuptake inhibitors (SSRIs) have become the leading class of antidepressants throughout the world. The efficacy and safety of SSRIs in the treatment of depression has been demonstrated in several clinical trials. With respect to safety, the studies show an advantage for the SSRIs over the older antidepressants. If the prescribing physicians are to make a well-founded judgement in their choice of drug factors like efficacy, safety, quality of life, and health economics must be taken into consideration. The primary aim of this study is to compare the efficacy of escitalopram with that of the serotonin norepinephrine reuptake inhibitors (SNRIs) duloxetine in the treatment of MDD.

ELIGIBILITY:
Inclusion Criteria:

* The patient suffers from a primary diagnosis of MDD according to DSM-IV-TR criteria (classification code 296.xx; current episode assessed using the MINI)
* The patient has a MADRS total score >=26 and a CGI-S score >=4 at the Baseline Visit

Exclusion Criteria:

* Any current psychiatric disorder other than MDD as defined in the DSM-IV TR
* Female patients of childbearing potential who are not using effective contraception
* Use of any psychoactive medication 2 weeks prior to screening and during the study

Other protocol-defined inclusion and exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2005-09; Primary Completion 2006-09 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
To compare the efficacy of escitalopram with that of duloxetine in outpatients with Major Depressive Disorder (MDD) as assessed by change in Montgomery-Åsberg Depression Rating Scale (MADRS) total score at the end of 24 weeks | 24 weeks

SECONDARY OUTCOMES:
To compare the efficacy of escitalopram with that of duloxetine per visit over the 24-week study period in outpatients with MDD. | Up to 24 weeks
  Secondary efficacy endpoints will be based on the MADRS, the Hamilton Depression Rating Scale (HAM-D17), the Hamilton Rating Scale for Anxiety (HAM-A), the CGI-S, the CGI-I and the Sheehan Disability Scale (SDS), Remission (MADRS<=12) and response (>=50% decrease from baseline in MADRS).
To compare the tolerability and safety of escitalopram with that of duloxetine over the 24-week study period in outpatients with MDD. | Up to 24 weeks
  Adverse events, clinical safety laboratory tests, vital signs
To evaluate the discontinuation emergent signs and symptoms during and after taper-down treatment with escitalopram or duloxetine after 24 weeks of treatment assessed by the Discontinuation Emergent Signs and Symptoms Scale (DESS). | Up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com

REFERENCES:
- [Result] Wade A, Gembert K, Florea I. A comparative study of the efficacy of acute and continuation treatment with escitalopram versus duloxetine in patients with major depressive disorder. Curr Med Res Opin. 2007 Jul;23(7):1605-14. doi: 10.1185/030079907x210732. PMID 17559755
- Available data/document: EMA EudraCT Results: 2004-005069-39 — https://www.clinicaltrialsregister.eu/ctr-search/trial/2004-005069-39/results